CLINICAL TRIAL: NCT01311804
Title: An Open Label,Multicentre, Randomized Trial to Determine the Efficacy of Periarticular Parecoxib Sodium In A Multimodal Cocktail vs Intravenous Parecoxib Sodium for Pain Management in Total Knee Arthroplasty
Brief Title: An Efficacy and Safety Study of Periarticular Parecoxib Sodium for Pain Management in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Dr. Yeap Ewe Juan, Name/Official Title: Dr. Yeap Ewe Juan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-2010; Ministry of Health (Other Grant/Funding Number: MOH)
Record Dates: First submitted 2011-03-03; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Unilateral Primary Osteoarthritis of Knee
MeSH Terms: interventions — parecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- periarticular parecoxib sodium (Experimental): patients will be given periarticular parecoxib sodium injection
  Interventions: Procedure: parecoxib sodium
- intravenous parecoxib sodium (Active Comparator): intravenous parecoxib sodium will be given during total knee arthroplasty
  Interventions: Procedure: parecoxib sodium

INTERVENTIONS:
Procedure: parecoxib sodium — periarticular parecoxib sodium injection will be given during total knee arthroplasty
  Other Names: dynastat
  Arms: periarticular parecoxib sodium
Procedure: parecoxib sodium — intravenous parecoxib sodium during total knee arthroplasty
  Other Names: dynastat
  Arms: intravenous parecoxib sodium

SUMMARY:
Primary Research Objective:

The primary objective of this study is to determine efficacy of periarticular parecoxib sodium in a multimodal cocktail versus intravenous parecoxib injections for pain management in total knee arthroplasty

Secondary Research Objective:

* To determine if perioperative use of parecoxib sodium was associated with improved clinical outcomes
* To evaluate the safety, in terms of adverse events; serious adverse events and tolerability of parecoxib sodium in periarticular injections in a multimodal cocktail

DETAILED DESCRIPTION:
This is a multi-center, open label, parallel randomized trial designed to evaluate the efficacy and safety of periarticular parecoxib sodium compared to intravenous parecoxib sodium.

125 patients with primary knee osteoarthritis from 4 participating sites who meet inclusion/exclusion criteria will be enrolled into the trial. After initial screening, patients will attend clinic for baseline examination. Subjects will then randomly allocated to periarticular parecoxib sodium or intravenous sodium in ratio of 1:1. patients are observed at post-operative 6, 12, 24 hours, subsequently daily for 4 days and finally at 2 week follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary knee osteoarthritis on treatment and planned for unilateral total knee arthroplasty and on spinal/general anesthesia
* Subjects age more than 50 and less than 85 years
* Patients with body weight at least 50 kg and not more than 50%above ideal body weight
* Written informed consent obtained from patient or guardian

Exclusion Criteria:

* Female patients who are attempting to conceive/pregnant
* Known allergy or hypersensitivity to cocktail regime or to COX-2 inhibitors
* History of bleeding disorders or coagulation defect
* Patients with abnormal liver profile
* Patients with history of stroke or major neurological defect
* Patients with neuropathic pain/sensory disorder
* Patients with peptic ulceration or anticoagulant use within 1 month
* History of previous major knee surgery/trauma
* Patients with renal insufficiency
* History of revision total knee arthroplasty
* Patients with knee deformity > 20 degrees
* Patients planned for bilateral knee arthroplasty during the same setting
* Patients with significant bone loss requiring augmentation
* Patients with history of using NSAIDs 24 hours before the surgery

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Post operative pain control | 4 days
  Post operative pain control( Visual Analogue Scale) with 0 corresponding to "no pain" and 10 to" the worst imaginable pain". Pain will be measured 1st 6 hours, 12 hours, 24 hours and daily for 4 days.

SECONDARY OUTCOMES:
Number and duration of adverse events | 4 days
  * Morphine consumption
  * Metochlopromide usage during the 4 days
  * Lactulose usage during the 4 days
  * Range of motion measured by physiotherapist at 24 hours and daily for 4 days
  * time to single leg raise
  * time to ambulation

CONTACTS AND LOCATIONS:
Overall Officials: Yeap Ewe Juan, Principal Investigator — MOH Malaysia
Locations (1):
- Hospital Tuanku Fauziah, Kangar, Perlis, Malaysia